CLINICAL TRIAL: NCT02435095
Title: Are Antipsychotics Neurotoxic or Neuroprotective? A Long-term Comparison of Two Treatment Strategies
Brief Title: Antipsychotic Induced Structural and Functional Brain Changes
Acronym: APIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow patient recruitment, low patient-commpliance, high dropout rates,
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-082
Record Dates: First submitted 2015-04-14; First posted 2015-05-06 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Maintenance treatment, Intermittent treatment; Brain volume; Antipsychotics
MeSH Terms: conditions — Schizophrenia | interventions — Opiate Substitution Treatment; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance treatment (Control) (Active Comparator): 287 female and male patients with schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) will be directed randomly to the maintenance treatment group (control). Patients will be treated according to the current clinical standard of long-term maintenance antipsychotic treatment. Study related procedures include safety assessments (physical examination, questionaires), laboratory assessments (blood sampling, urine analysis), efficacy assessments (questionaires) and volumetric Magnetic Resonance Imaging (structural MRI incl. volumetry). Study procedures are the same for both study groups (control/experimental).
  Interventions: Drug: Maintenance treatment
- Intermittent Treatment (Experimental) (Experimental): 287 female and male patients with schizophrenia according to DSM-V will be directed randomly to the intermittent treatment group (experimental). Patients directed to this group will be tapered off medication.
  Study related procedures include safety assessments (physical examination, questionaires), laboratory assessments (blood sampling, urine analysis), efficacy assessments (questionaires) and volumetric Magnetic Resonance Imaging (structural MRI incl. volumetry). Study procedures are the same for both study groups (control/experimental).
  Interventions: Drug: Intermittent treatment

INTERVENTIONS:
Drug: Maintenance treatment — Treatment with antipsychotic drug (either second-generation antipsychotics or low-dose first generation antipsychotics) for at least 12 months.
  All antipsychotics approved in Germany are permitted (amisulpride, aripiprazole, benperidol, bromperidol, chlorprothixene, clozapine, flupentixole, fluphenazine, fluspirilene, haloperidol, levomepromazine, loxapine, lurasidone, melperone, olanzapine, paliperidone, perazine, perphenazine, pimozide, pipamperone, prothipendyl, quetiapine, risperidone, sertindole, sulpiride, thioridazine, ziprasidone, zuclopenthixole).
  Other Names: Antipsychotics
  Arms: Maintenance treatment (Control)
Drug: Intermittent treatment — Treatment with antipsychotic drug (either second-generation antipsychotics or low-dose first generation antipsychotics) only for first episode of schizophrenia, tapering-off medication after remission of positive symptoms, reinstatement of treatment only in case of recurrence of positive symptoms.
  All antipsychotics approved in Germany are permitted (amisulpride, aripiprazole, benperidol, bromperidol, chlorprothixene, clozapine, flupentixole, fluphenazine, fluspirilene, haloperidol, levomepromazine, loxapine, lurasidone, melperone, olanzapine, paliperidone, perazine, perphenazine, pimozide, pipamperone, prothipendyl, quetiapine, risperidone, sertindole, sulpiride, thioridazine, ziprasidone, zuclopenthixole).
  Other Names: Antipsychotics
  Arms: Intermittent Treatment (Experimental)

SUMMARY:
Continuation of antipsychotic drug treatment for at least 12 months after remission of the first psychotic episode represents the gold clinical standard, and it is recommended by all international treatment guidelines. Numerous studies have shown that the risk of relapse is significantly increased, if drug treatment is terminated prematurely. However, only a minority of patients achieve functional remission, even if they fully comply with treatment. Long-term adverse effects of the currently available drugs, specifically brain grey matter loss and development of supersensitivity psychosis, might outweigh their benefits. Thus, the current standard of long-term maintenance antipsychotic treatment, which has the primary goal of relapse prevention, has to be questioned. Here the investigators hypothesize that intermittent treatment (experimental) with antipsychotics, which is directed exclusively against the positive symptoms of Schizophrenia, is associated with less loss in total grey matter volume than maintenance treatment (control). Furthermore, the investigators hypothesise that this targeted treatment approach is associated with better functional outcome (fewer negative symptoms, better cognitive performance, better quality of life) than continuous antipsychotic treatment,although the latter is initially associated with fewer relapses.The aim of the present study is to compare two different drug therapies -maintenance therapy versus on-demand, intermittent therapy- in terms of their treatment's success and the structural changes in the brain.

DETAILED DESCRIPTION:
Patients with diagnosis of schizophrenia according to DSM-5 admitted to a hospital participating in the consortium will undergo magnetic resonance imaging (MRI) as soon as possible after admission. Ideally, this procedure is performed before initiation of antipsychotic treatment (benzodiazepines are allowed). If not possible for clinical reasons, antipsychotic treatment will be started and the MRI will be acquired within three days of initiation of drug treatment. The choice of the antipsychotic will be made by the treating physician. All approved antipsychotics are permitted, including first-generation antipsychotics such as haloperidol or flupenthixol. This is based on the recommendation of the British NICE guidelines: "In nine randomized controlled trials (RCTs) with a total of 1,801 participants with first-episode or early schizophrenia (including people with a recent onset of schizophrenia and people who have never been treated with antipsychotic medication), the evidence suggested there were no clinically significant differences in efficacy between the antipsychotic drugs examined." (NICE 2009, p. 105). However, since second-generation antipsychotics (SGA) are now considered first-line treatment for schizophrenia according to the German S3 guideline, it can be assumed that more than 80% of all patients will be treated with an SGA.

As soon as positive symptoms are sufficiently controlled, medication will be completely tapered off within four weeks. Sufficient control of positive symptoms will defined as follows: "delusions" (Positive and Negative Syndrome Scale (PANSS) item 1), "hallucinatory behaviour" (PANSS item 3), and "suspiciousness/persecution" (PANSS item 6) have to be "absent" or "mild" (scores 1 or 2). The PANSS Positive score (7 items) must not be above 18. Patients in the experimental group who will not reach remission according to this definition will be switched to another antipsychotic according to clinical standards. Tapering of medication might be considered at a later time-point. Patients who cannot be tapered off medication will be treated with the lowest possible dose.

Treatment of subsequent exacerbations / psychotic relapses will follow the same rules.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of schizophrenia according to DSM-5
* Age 18-65 years
* Written declaration of consent
* Subjects being contractually and mentally capable to attend the medical staffs' orders.
* MRI capability

Exclusion Criteria:

* Relevant somatic diseases, which could have an impact on the conduct of the study based on clinical judgement of the treating physician (e.g. epilepsy, cancer)
* Prior insufficiently documented drug therapy with antipsychotics
* Magnetic metals in and on the body, cardiac pacemakers and body piercings.
* Pregnancy or lactation
* Hospitalization of the patient ordered by the court or public authorities
* Relationship of dependence or employment to sponsor or investigator
* Simultaneous participation in another clinical trial (participation in an APIC subproject excluded)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-05; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Total grey matter volume | over 12 months
  change in total grey matter volume

SECONDARY OUTCOMES:
Grey matter volume (hippocampus, prefrontal cortex) | after 6 and 24 months
  change of volume
Assessment of safety as assessed with the following instrument: EPS | after 6 and 12 months
  Extrapyramidal symptom scale (EPS)
Assessment of safety as assessed with the following instrument: BARS | after 6 and 12 months
  Barnes Akathisia Rating Scale (BARS)
Assessment of safety as assessed with the following instrument: Arizona Scale | after 6 and 12 months
  Sexual function (Arizona Scale)
Global assessment of safety as assessed with laboratory values | after 6 and 12 months
  Metabolic side effects (Body mass index, HbA1c, Glucose, Cholesterol, Triglycerides)
Cognition | after 6 and 12 months
  Brief Assessment of Cognition in Schizophrenia (BACS)
Quality of life | after 6 and 12 months
  Short Form-36 Health Survey (SF-36), Global Assessment of Functioning Scale (GAF), visual analogue scales
Psychopathology as assessed with the PANSS | after 6 and 12 months
  Positive and Negative Syndrome Scale (PANSS)
Psychopathology as assessed with the CGI | after 6 and 12 months
  Clinical Global Impression (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mathiak, Univ.-Prof. Dr. Dr., Principal Investigator — Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital RWTH Aachen, Germany
Locations (11):
- Germany (11):
  - RWTH University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Alexianer Aachen GmbH, Aachen
  - Zentrum für Neurologie und Seelische Gesundheit im Kapuziner Karree Aachen, Aachen
  - LVR Klinik Bonn, Bonn
  - LVR Klinik Düren, Düren
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie der Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - LVR Klinik Essen, Essen
  - ViaNobis Gangelt, Gangelt
  - Klinik Königshof (Abteilung für Allgemeine Psychiatrie), Krefeld
  - LVR Klinik Langenfeld, Langenfeld
  - LVR Klinik Viersen, Viersen